CLINICAL TRIAL: NCT02479334
Title: Acute Effects of Spices on Pathways Associated With Glucose Homeostasis, Oxidative Stress and Inflammation in Healthy Subjects - Molecular Insights Through Transcriptomics of Peripheral Blood Mononuclear Cells (PBMC)
Brief Title: Acute Effects of Spices on Pathways Associated With Glucose Homeostasis and Inflammation on PBMCs of Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Food for Health Science Centre, Lund University (Unknown)
Responsible Party: Principal Investigator, Elin Östman, Assoc. Prof. PhD., Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LUND-AFC-STAGE3-SPICENUTROMICS
Record Dates: First submitted 2015-03-30; First posted 2015-06-24 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Spices; Functional food; Cardiometabolic risk; Metabolic syndrome; Inflammation; Peripheral blood mononuclear cell; Acute
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fat challenge breakfast (Placebo Comparator): 200 ml control drink (non-energy flavored water) and high fat breakfast (% Energy Carbohydrate:Fat:Prot / 20:60:20), acute study / one time administration
  Interventions: Other: Fat challenge breakfast
- Fat challenge breakfast+spices (Experimental): 200 ml spices drink (non-energy flavored water + spices extract) and high fat breakfast (% Energy Carbohydrate:Fat:Prot / 20:60:20), acute study / one time administration
  Interventions: Other: Fat challenge breakfast+spices
- Carbohydrate challenge breakfast (Placebo Comparator): 200 ml control drink (non-energy flavored water) and high carbohydrate breakfast (% Energy Carbohydrate:Fat:Prot / 60:20:20), acute study / one time administration
  Interventions: Other: Carbohydrate challenge breakfast
- Carbohydrate challenge breakfast+spices (Experimental): 200 ml spices drink (non-energy flavored water + spices extract) and high carbohydrate breakfast (% Energy Carbohydrate:Fat:Prot / 60:20:20), acute study / one time administration
  Interventions: Other: Carbohydrate challenge breakfast+spices

INTERVENTIONS:
Other: Fat challenge breakfast — In this intervention, subjects are asked to consume 200 ml control drinks (non-energy flavored water). Following 10 min. beverage consumption, subjects will be given standardized high fat breakfast corresponding to % Energy of Carbohydrate:Fat:Prot / 20:60:20
  Arms: Fat challenge breakfast
Other: Fat challenge breakfast+spices — In this intervention, subjects are asked to consume 200 ml spices drinks (non-energy flavored water + spices extract). Following 10 min. beverage consumption, subjects will be given standardized high fat breakfast corresponding to % Energy of Carbohydrate:Fat:Prot / 20:60:20
  Arms: Fat challenge breakfast+spices
Other: Carbohydrate challenge breakfast — In this intervention, subjects are asked to consume 200 ml control drinks (non-energy flavored water). Following 10 min. beverage consumption, subjects will be given standardized high carbohydrate breakfast corresponding to % Energy of Carbohydrate:Fat:Prot / 60:20:20
  Arms: Carbohydrate challenge breakfast
Other: Carbohydrate challenge breakfast+spices — In this intervention, subjects are asked to consume 200 ml spices drinks (non-energy flavored water + spices extract). Following 10 min. beverage consumption, subjects will be given standardized high carbohydrate breakfast corresponding to % Energy of Carbohydrate:Fat:Prot / 60:20:20
  Arms: Carbohydrate challenge breakfast+spices

SUMMARY:
This study aims to investigate the effect of spices on gene expression of pathways associated with glucose homeostasis, oxidative stress and inflammation, in the postprandial phase in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* BMI 20-28 kg/m2
* Must be able to accept spices
* Agreed and signed informed consent

Exclusion Criteria:

* Below 18 years old
* Uncomfortable speaking English and/or difficulties in understanding spoken English
* Smoking or using snuss
* Vegetarian or vegan
* Stressed by venous blood sampling or previous experience of being difficult to be cannulated
* Receiving any drug treatment that may influence the study outcomes
* Pregnancy or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (0 hr) in untargeted PBMC gene expression profile at 2 hr and 4 hr | Prior to the initial intervention at 0 hr and after intervention at 2 hr and 4 hr.
  The venous blood samples will be taken for isolation of peripheral blood mononuclear cells. Extracted total RNA will then be used for running RNA-seq/whole-transcriptome shotgun sequencing (Illumina, San Diego, CA, USA)

SECONDARY OUTCOMES:
Subjective appetite ratings using standard subjective 100 mm VAS | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  Appetite will be assessed using standard subjective 100 mm VAS (visual analogue scale) at time intervals throughout each visit
Metabolic biomarkers | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  The capillary blood samples will be taken for blood glucose analysis. The venous blood samples will be taken for further assessment of insulin, triacylglycerol, NEFA and inflammatory biomarkers (i.e. IL-6, IL-8, CRP)
Metabolite profile | Prior to the initial intervention at 0 min and after intervention at 15, 30, 45, 60, 90, 120, 180 and 240 min.
  Metabolite profile will be analyzed using Liquid Chromatography-Mass Spectrometry based methods

CONTACTS AND LOCATIONS:
Overall Officials: Yoghatama Cindya Zanzer, MSc, Study Chair — Lund University; Elin Östman, PhD, Principal Investigator — Lund University
Locations (1):
- Food for Health Laboratory - Lund University, Lund, Skåne County, Sweden